CLINICAL TRIAL: NCT06229899
Title: Can Follistatin Levels Help Distinguish Between Metabolically Healthy and Unhealthy Obese Individuals
Brief Title: Follistatin Levels in Metabolically Healthy and Unhealthy Obese Individuals
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: Metabolic health-Follistatin
Record Dates: First submitted 2024-01-15; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples for follistatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metabolically healthy individuals with obesity: Individuals with BMI ≥30 , those without criteria of metabolic syndrome other than an increase in waist circumference (blood pressure ≥130/85 mmHg, fasting blood sugar ≥100 mg/dl, triglycerides ≥150 mg/dl, HDL-cholesterol <40 mg/dl in men and <50 mg/dl in women) and without prediabetes
  Interventions: Diagnostic Test: Serum follistatin levels
- metabolically unhealthy individuals with obesity: Individuals with BMI ≥30 , and have one of the followings: blood pressure ≥130/85 mmHg, fasting blood sugar ≥100 mg/dl, triglycerides ≥150 mg/dl, HDL-cholesterol <40 mg/dl in men and <50 mg/dl in women
  Interventions: Diagnostic Test: Serum follistatin levels

INTERVENTIONS:
Diagnostic Test: Serum follistatin levels — blood samples are taken

SUMMARY:
There is no clear boundary on which obese individuals should be considered metabolically healthy and which should be considered metabolically unhealthy. It is also not very clear whether the individuals who are considered metabolically healthy will remain healthy in the future. The objective of this study was to assess potential disparities in serum follistatin levels between these two distinct groups. Furthermore, the study sought to investigate whether this disparity could serve as a reliable indicator for distinguishing between metabolically healthy and unhealthy obese individuals.

DETAILED DESCRIPTION:
Individuals with similar body mass indexes may have different metabolic health and cardiovascular risks. Research shows that some individuals with comparable body mass index (BMI) are metabolically healthy and have a lower risk of cardiovascular issues, while others are metabolically unhealthy and have a higher risk. Studies indicate that the lifestyles of metabolically healthy and unhealthy obese individuals, such as diet, physical activity, and sleep patterns, do not differ significantly, even though the individuals have similar levels of total or subcutaneous adiposity. However, it has been shown that metabolically healthy obese individuals tend to have lower levels of visceral adiposity compared to unhealthy ones.

Patients with BMI≥30, who applied to the internal medicine clinic, were included in the study. Among these patients, those without criteria of metabolic syndrome other than an increase in waist circumference (blood pressure ≥130/85 mmHg, fasting blood sugar ≥100 mg/dl, triglycerides ≥150 mg/dl, HDL-cholesterol <40 mg/dl in men and <50 mg/dl in women) and without prediabetes were defined as metabolically healthy obese individuals. Those with at least 1 metabolic syndrome criterion other than an increase in waist circumference were classified as metabolically unhealthy obese individuals. The participants' fasting blood sugar levels, HbA1c levels, insulin levels, lipid panel results, liver enzymes levels,urea levels, creatinine levels, whole blood count, and thyroid hormones were examined. Anthropometric measurements including height,weight and waist circumference were also taken for each individual.

Participants were then invited back to repeat follistatin levels.

ELIGIBILITY:
Inclusion Criteria:

* Having given consent to the study
* Being over 18 years of age
* Being under 60 years of age
* Body mass index >=30 kg/m2

Exclusion Criteria:

* Antidiabetic medication usage
* obesity surgery
* Antihypertensive medication usage
* Those receiving lipid-lowering therapy
* Pregnant women
* Those with hypo/hyperthyroidism
* Steroid use
* Benign/malignant tumors
* Advanced liver disease
* Secondary causes of obesity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals between 18-60 years old, with a BMI of ≥ 30, who are not using any medication or have any disease that may effect their glycemia, lipid profiles or blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
relation between follistatin and metabolically healthy and unhealthy obesity | baseline
  This study aims to examine the correlation between follistatin levels and both metabolically healthy and unhealthy individuals with obesity
threshold for follistatin in metabolic evaluation of obesity | baseline
  The establishment of a threshold value for follistatin levels in assessing metabolic health in obese individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe N Erbakan, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Research and TRaining Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Research and TRaining Hospital, Istanbul, Turkey (Türkiye)